CLINICAL TRIAL: NCT07307859
Title: Effect of Pain Neuroscience Education Combined With Lumbar Stabilization Exercises on Disability and Kinesiophobia Among Patients With Chronic Low Back Pain
Brief Title: Pain Neuroscience Education Combined With Lumbar Stabilization Exercises on Disability and Kinesiophobia Among Patients With Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mosab ALdabbas, Assistant Professor at Al Azhar University ,Palestine, Gaza, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Al Azhar University , Gaza
Record Dates: First submitted 2025-12-05; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low Back Pain
Keywords: pain neuroscience; lumbar stabilization; disability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar Stabilization Exercises (Active Comparator): Standard Lumbar Stabilization Exercise Program A physiotherapy program focused solely on core and trunk stabilization exercises without additional educational components.
  Interventions: Other: Control Group - Lumbar Stabilization Exercises Only
- Lumbar Stabilization Exercises Plus Pain Neuroscience Education (Experimental): Lumbar Stabilization Program Integrated with Weekly Pain Neuroscience Education Sessions A combined intervention including trunk stabilization exercises supported by once-weekly educational sessions addressing pain mechanisms and fear-avoidance beliefs.
  Interventions: Other: Experimental Group - Lumbar Stabilization Exercises + PNE

INTERVENTIONS:
Other: Experimental Group - Lumbar Stabilization Exercises + PNE — Experimental Group - Lumbar Stabilization Exercises + PNE
  1. Lumbar Stabilization Exercises (LSE)
     Frequency: 3 supervised sessions per week for 8 weeks
     → Total 24 supervised LSE sessions
     Session duration: 45-60 minutes
     Structure each session:
     Warm-up (5-10 min)
     Core stabilization program (30-40 min)
     Cool-down (5-10 min)
     Progression: Exercises will advance weekly from basic motor control to high-level functional stabilization (details below).
     Home program: 1 additional short home session weekly (basic LSE).
     Monitoring: VAS before and after each session. Exercises will be modified if pain rises >2 VAS points.
     Adherence: Attendance logs
  2. Pain Neuroscience Education (PNE)
  Frequency: Once per week (included within one of the 3 weekly sessions)
  → Total 8 PNE sessions
  Duration: 30-40 minutes
  Format: Small group (≤5) or one-on-one
  Methods: Metaphors, storytelling, diagrams, role-play, Arabic handouts
  Learning evaluation: Mini-quizzes, reflective journaling, i
  Arms: Lumbar Stabilization Exercises Plus Pain Neuroscience Education
Other: Control Group - Lumbar Stabilization Exercises Only — Lumbar Stabilization Exercises (LSE)
  Frequency: 3 supervised sessions per week for 8 weeks
  → Total 24 supervised LSE sessions
  Session duration: 45-60 minutes
  Structure: Identical warm-up, core program, and cool-down as the experimental group.
  Progression: Identical 8-week exercise progression.
  Home program: 1 basic LSE home session weekly (same as experimental group).
  Communication: Therapists will not provide pain education or discuss pain science concepts.
  Adherence: Attendance logs and SMS reminders identical to the experimental group.
  Arms: Lumbar Stabilization Exercises

SUMMARY:
This study will investigate the effect of adding Pain Neuroscience Education (PNE) to a standard lumbar stabilization exercise program on disability and kinesiophobia among patients with chronic low back pain in the Gaza Strip. Participants will be randomly assigned into two groups:

Control group - will receive lumbar stabilization exercises only.

Experimental group - will receive lumbar stabilization exercises in addition to PNE delivered once weekly for 8 sessions.

Both groups will undergo an 8-week intervention, and outcome measures will be collected at baseline, post-intervention (8 weeks), and at a follow-up assessment (16 weeks) to evaluate the persistence of treatment effects. It is expected that the experimental group will show greater improvements in disability and kinesiophobia compared with the control group, indicating that integrating PNE with stabilization exercises may provide enhanced and sustained benefits for patients with chronic low back pain.

DETAILED DESCRIPTION:
This study will explore whether integrating Pain Neuroscience Education (PNE) with a lumbar stabilization exercise program can produce superior clinical outcomes for individuals with chronic low back pain. The intervention will be delivered over eight weeks, with both groups participating in supervised lumbar stabilization sessions. The experimental group will additionally receive weekly PNE sessions designed to improve pain understanding, modify unhelpful beliefs, and reduce fear-avoidance behaviors.

PNE sessions will focus on explaining the neurophysiological mechanisms of chronic pain, emphasizing concepts such as central sensitization, the protective nature of pain, and the role of thoughts, emotions, and movement in pain modulation. The lumbar stabilization exercises will aim to improve trunk control, enhance spinal stability, and promote functional movement patterns.

Participants will be assessed at baseline, after completion of the intervention period, and again at a later follow-up to examine the sustainability of treatment effects. The study is expected to provide evidence on whether combining educational and physical interventions yields greater improvements in disability and kinesiophobia compared with stabilization exercises alone. This information may support future clinical decision-making and contribute to improving physiotherapy services for patients with chronic low back pain in the Gaza Strip.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 25to 50 years.
* CLBP lasting for more than 12 weeks.

Exclusion Criteria:

* History of spinal surgery or fractures.
* Presence of neurological problems.
* Inflammatory conditions, including radiculopathy.
* Pregnancy.
* Body mass index (BMI) ≥ 30.
* Chronic systemic diseases or conditions requiring regular use of strong analgesics or opioids, which may interfere with intervention outcomes.
* Significant visual or hearing impairments.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | Time Frame: Baseline (pre-intervention), immediately post-intervention at 8 weeks, and follow-up at 8 weeks post-intervention (16 weeks from baseline).
  Oswestry Disability Index (ODI) The ODI is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each topic category will be followed by six statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5, with the first statement being zero and indicating the least amount of disability. The last statement will score5, showing the most severe 18 disability. The scores for all questions answered are summed and then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability, and
Tampa Scale for Kinesiophobia (TSK) | Time Frame: Baseline (pre-intervention), immediately post-intervention at 8 weeks, and follow-up at 8 weeks post-intervention (16 weeks from baseline).
  The Tampa Scale for Kinesiophobia (TSK) is a widely used, validated self-report questionnaire designed to assess fear of movement and fear-avoidance beliefs in individuals with musculoskeletal pain, particularly chronic low back pain. The scale measures the degree to which a person fears that movement or physical activity may cause pain or lead to reinjury.
  The TSK consists of 17 items, each rated on a 4-point Likert scale ranging from:
  1. = Strongly disagree
  2. = Disagree
  3. = Agree
  4. = Strongly agree
  The total score ranges from 17 to 68, with higher scores indicating greater levels of kinesiophobia, meaning stronger fear-avoidance behavior, increased movement-related fear, and greater concern about physical activity causing harm.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Time Frame: Baseline (pre-intervention), immediately post-intervention at 8 weeks, and follow-up at 8 weeks post-intervention (16 weeks from baseline).
  The Visual Analog Scale (VAS) is a widely used and validated tool for assessing subjective pain intensity in both acute and chronic pain conditions. It is simple, sensitive, and responsive to changes in pain, making it suitable for clinical trials and re

IPD SHARING:
Plan to Share IPD: No